CLINICAL TRIAL: NCT05411562
Title: On-Demand Point-of-Care SARS-CoV-2 Genomic Sequencing to Support Nosocomial Outbreak Investigations: A Prospective Molecular Epidemiology Study in Montreal
Brief Title: COVID-19 Genomic Sequencing for Nosocomial Outbreak Investigations
Acronym: NOSO-COVID
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 20.270
Record Dates: First submitted 2022-06-02; First posted 2022-06-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; Molecular Sequence Variation; Nosocomial Infection
MeSH Terms: conditions — COVID-19; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs from patients and healthcare workers. Primary samples that are positive on PCR or SARS-CoV-2 are retained.

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 genomic sequencing — SARS-CoV-2 viral genomic sequencing and phylogenetic analyses

SUMMARY:
This is a tertiary care hospital-based prospective molecular epidemiology study in Montreal, Canada. When nosocomial transmission was suspected by local infection control teams' investigations, SARS-CoV-2 viral genomic sequencing was performed locally for all putative outbreak cases and contemporary controls. Molecular and conventional epidemiology data were confronted in real time to improve understanding of COVID-19 transmission and reinforce or adapt prevention measures.

DETAILED DESCRIPTION:
This study will include infected healthcare workers (HCW) and patients for whom a nosocomial infection in CHUM is suspected. The CHUM laboratory is responsible for COVID-19 diagnostic testing in all eligible HCW and patients. After initial diagnosis on standard PCR testing, samples are maintained at -80. Viral RNA is extracted and next-generation sequencing of the viral genome is performed using Nanopore long read sequencing platform. Preliminary data suggest that SARS-CoV-2 has a "molecular clock" of 2 single nucleotide polymorphism (SNP) per month. The analysis and between-isolate comparaison of those SNP among epidemiologically related cases will allow to support or refute the hypothesis of person to person nosocomial transmission. All infected patients will be matched 1:1 with contemporary community cases to provide a viral genome back catalog and better contextualize molecular epidemiology analyses. Molecular clusters will be reported to infection prevention and control teams and resulting interventions will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the institution during the study period
* Healthcare workers in the institution during the study period

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthcare workers in the institution during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Outbreak control measures improvement | Through study completion, an average of 2 years
  Collaborative (infection control and molecular epidemiology teams) resolution of putative outbreaks. Transmission is either refuted or further supported by molecular analyses. Additional investigation efforts are discontinued or necessary corrective measures are implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Grandjean Lapierre, MD MSc FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Viral genomic sequences from all participants are to be deposited on GenBank.

REFERENCES:
- [Derived] Benoit P, Jolicoeur G, Point F, Soucy C, Normand K, Morency-Potvin P, Gagnon S, Kaufmann DE, Tremblay C, Coutlee F, Harrigan PR, Hardy I, Smith M, Savard P, Grandjean Lapierre S. On-demand, hospital-based, severe acute respiratory coronavirus virus 2 (SARS-CoV-2) genomic epidemiology to support nosocomial outbreak investigations: A prospective molecular epidemiology study. Antimicrob Steward Healthc Epidemiol. 2023 Mar 8;3(1):e45. doi: 10.1017/ash.2023.119. eCollection 2023. PMID 36960087